CLINICAL TRIAL: NCT02980302
Title: Development of the Tool " iPSC " (Induced Pluripotent Stem Cells) for the Functional Study of Mutations Responsible for Mental Retardation - Application to Familial Study of MYT1L Gene Mutations
Brief Title: Development of the Tool " iPSC " for the Functional Study of Mutations Responsible for Mental Retardation
Acronym: Rementips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC14.181
Record Dates: First submitted 2016-07-28; First posted 2016-12-02 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Intellectual Deficiency; Asymptomatic Carrier of the Mutation of the Gene MYT1L; Healthy Volunteers
Keywords: Mental retardation MR; IQ; Mutation; Gene MYT1L

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patient (Other)
  Interventions: Procedure: Cutaneous biopsy
- Asymptomatic carrier (Other): Father of the patient : asymptomatic carrier of the same mutation
  Interventions: Procedure: Cutaneous biopsy
- Two control patients (Other)
  Interventions: Procedure: Cutaneous biopsy

INTERVENTIONS:
Procedure: Cutaneous biopsy — Under local anesthesia

SUMMARY:
According to the World Health Organization (WHO), mental retardation (MR) is defined by an intelligence quotient (IQ) < 70 and touches between 1 to 3 % of the general population. Profound mental retardation (QI <25), severe (IQ: 25-40) and moderate (QI : 40-50) have a prevalence of 0,3-0,5% while the prevalence of mild MR, defined by an IQ between 50 and 70 is evaluated to about 1,5 %.

The origin of MR can be infectious, toxic, traumatic, genetic or environmental. genetic causes of MR gather the number and structure anomalies of the chromosomes, the genomic microreorganization, monogenic diseases and more rarely other non Mendelian-inherited anomalies like print or epigenetic anomalies, mutations of the mitochondrial genome etc... Genetic causes represents 50% of moderate to severe, whereas environmental factors (malnutrition, cultural deprivation,...) plays an important role in mild MR.

The main goal of this study is to get an innovative tool (neuronal distinction of iPSC) that wil allow to study the functionnal impact of mutations uppon genes probably involved in MR like MYT1L. The main criteria associated to characterisation of the tool by the trial is the study of the pluripotency of iPSC obtained and to highlight the mutation of the gene MYT1L in the iPSC.

Neurons from the iPSC of the patient and his father du patient wille also be morphologically characterised, but also thanks to the expression of specifically neurals genes.

Characteristics of iPSC and neurons from d'iPSC with MYT1L mutation will be compared among the patient and his father, in relation with the same cells coming from the two witnesses.

ELIGIBILITY:
Inclusion Criteria :

* Patient with an intellectual deficiency and/or associated signs that received a chromosomic analysis by CGH-array revealing a variant of unknown signification involvingone or more genes candidates for mental retardation.
* Certificate of genetic genetic counselling and signed consent.
* Under 18 persons may be necessary because intellectual deficiency is often diagnosed before the adult age.
* Number of cases is very limited in this preliminary study and only one patient showing a rare mutation of MYT1L gene and his father ( asymptomatic carrier of the same mutation) will be study.
* Affiliation to a social security system

Exclusion Criteria :

* Persons mentionned L1121-5 to L1121-8 of CSP (all protected persons)
* Persons suffering from acute infections for the practice of cutaneous biopsy under local anesthesia.
* Persons showing an hemostasis disorder acquired or induced
* Persons sous traitement antiagrégant anticoagulant
* Persons with a mutation in th gene MYT1L

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
iPSC caracterization from human fibroblast with MYT1L mutation | Half an hour
  Skin sampling under local anesthesia. Evaluation of iPSC gene expression for their pluripotency.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Simon Jouk, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Bonnet C, Leheup B, Beri M, Philippe C, Gregoire MJ, Jonveaux P. Aberrant GRIA3 transcripts with multi-exon duplications in a family with X-linked mental retardation. Am J Med Genet A. 2009 Jun;149A(6):1280-9. doi: 10.1002/ajmg.a.32858. PMID 19449417
- [Background] Brosco JP, Mattingly M, Sanders LM. Impact of specific medical interventions on reducing the prevalence of mental retardation. Arch Pediatr Adolesc Med. 2006 Mar;160(3):302-9. doi: 10.1001/archpedi.160.3.302. PMID 16520451
- [Background] Chambers SM, Fasano CA, Papapetrou EP, Tomishima M, Sadelain M, Studer L. Highly efficient neural conversion of human ES and iPS cells by dual inhibition of SMAD signaling. Nat Biotechnol. 2009 Mar;27(3):275-80. doi: 10.1038/nbt.1529. Epub 2009 Mar 1. PMID 19252484
- [Background] Chanda S, Marro S, Wernig M, Sudhof TC. Neurons generated by direct conversion of fibroblasts reproduce synaptic phenotype caused by autism-associated neuroligin-3 mutation. Proc Natl Acad Sci U S A. 2013 Oct 8;110(41):16622-7. doi: 10.1073/pnas.1316240110. Epub 2013 Sep 17. PMID 24046374
- [Background] Chiurazzi P, Schwartz CE, Gecz J, Neri G. XLMR genes: update 2007. Eur J Hum Genet. 2008 Apr;16(4):422-34. doi: 10.1038/sj.ejhg.5201994. Epub 2008 Jan 16. PMID 18197188
- [Background] Chiyonobu T, Hayashi S, Kobayashi K, Morimoto M, Miyanomae Y, Nishimura A, Nishimoto A, Ito C, Imoto I, Sugimoto T, Jia Z, Inazawa J, Toda T. Partial tandem duplication of GRIA3 in a male with mental retardation. Am J Med Genet A. 2007 Jul 1;143A(13):1448-55. doi: 10.1002/ajmg.a.31798. PMID 17568425
- [Background] Cohn DM, Pagon RA, Hudgins L, Schwartz CE, Stevenson RE, Friez MJ. Partial ATRX gene duplication causes ATR-X syndrome. Am J Med Genet A. 2009 Oct;149A(10):2317-20. doi: 10.1002/ajmg.a.33006. No abstract available. PMID 19764021
- [Background] Doco-Fenzy M, Leroy C, Schneider A, Petit F, Delrue MA, Andrieux J, Perrin-Sabourin L, Landais E, Aboura A, Puechberty J, Girard M, Tournaire M, Sanchez E, Rooryck C, Ameil A, Goossens M, Jonveaux P, Lefort G, Taine L, Cailley D, Gaillard D, Leheup B, Sarda P, Genevieve D. Early-onset obesity and paternal 2pter deletion encompassing the ACP1, TMEM18, and MYT1L genes. Eur J Hum Genet. 2014 Apr;22(4):471-9. doi: 10.1038/ejhg.2013.189. Epub 2013 Oct 16. PMID 24129437
- [Background] Froyen G, Belet S, Martinez F, Santos-Reboucas CB, Declercq M, Verbeeck J, Donckers L, Berland S, Mayo S, Rosello M, Pimentel MM, Fintelman-Rodrigues N, Hovland R, Rodrigues dos Santos S, Raymond FL, Bose T, Corbett MA, Sheffield L, van Ravenswaaij-Arts CM, Dijkhuizen T, Coutton C, Satre V, Siu V, Marynen P. Copy-number gains of HUWE1 due to replication- and recombination-based rearrangements. Am J Hum Genet. 2012 Aug 10;91(2):252-64. doi: 10.1016/j.ajhg.2012.06.010. Epub 2012 Jul 26. PMID 22840365
- [Background] Kearney HM, Thorland EC, Brown KK, Quintero-Rivera F, South ST; Working Group of the American College of Medical Genetics Laboratory Quality Assurance Committee. American College of Medical Genetics standards and guidelines for interpretation and reporting of postnatal constitutional copy number variants. Genet Med. 2011 Jul;13(7):680-5. doi: 10.1097/GIM.0b013e3182217a3a. PMID 21681106
- [Background] Kleinjan DA, van Heyningen V. Long-range control of gene expression: emerging mechanisms and disruption in disease. Am J Hum Genet. 2005 Jan;76(1):8-32. doi: 10.1086/426833. Epub 2004 Nov 17. PMID 15549674
- [Background] Larson SA, Lakin KC, Anderson L, Kwak N, Lee JH, Anderson D. Prevalence of mental retardation and developmental disabilities: estimates from the 1994/1995 National Health Interview Survey Disability Supplements. Am J Ment Retard. 2001 May;106(3):231-52. PMID 11408960
- [Background] Lee C, Iafrate AJ, Brothman AR. Copy number variations and clinical cytogenetic diagnosis of constitutional disorders. Nat Genet. 2007 Jul;39(7 Suppl):S48-54. doi: 10.1038/ng2092. PMID 17597782
- [Background] Lujan E, Chanda S, Ahlenius H, Sudhof TC, Wernig M. Direct conversion of mouse fibroblasts to self-renewing, tripotent neural precursor cells. Proc Natl Acad Sci U S A. 2012 Feb 14;109(7):2527-32. doi: 10.1073/pnas.1121003109. Epub 2012 Jan 30. PMID 22308465
- [Background] McLaren J, Bryson SE. Review of recent epidemiological studies of mental retardation: prevalence, associated disorders, and etiology. Am J Ment Retard. 1987 Nov;92(3):243-54. PMID 3322329
- [Background] Raff ML, Craigen WJ, Smith LT, Keene DR, Byers PH. Partial COL1A2 gene duplication produces features of osteogenesis imperfecta and Ehlers-Danlos syndrome type VII. Hum Genet. 2000 Jan;106(1):19-28. doi: 10.1007/s004390051004. PMID 10982177
- [Background] Pang ZP, Yang N, Vierbuchen T, Ostermeier A, Fuentes DR, Yang TQ, Citri A, Sebastiano V, Marro S, Sudhof TC, Wernig M. Induction of human neuronal cells by defined transcription factors. Nature. 2011 May 26;476(7359):220-3. doi: 10.1038/nature10202. PMID 21617644
- [Background] Rodriguez-Revenga L, Mila M, Rosenberg C, Lamb A, Lee C. Structural variation in the human genome: the impact of copy number variants on clinical diagnosis. Genet Med. 2007 Sep;9(9):600-6. doi: 10.1097/gim.0b013e318149e1e3. PMID 17873648
- [Background] Rooryck Thambo C. Analyse de réarrangements génomiques chez des patients atteints d'anomalies du développement embryonnaire. Retard mental et malformations multiples congénitales ; Spectre oculo-auriculo-vertébral. 2009. Thèse de science n°1675. Ecole doctorale des sciences de la vie et de la santé, université Bordeaux 2.
- [Background] Shimojima K, Inoue T, Imai Y, Arai Y, Komoike Y, Sugawara M, Fujita T, Ideguchi H, Yasumoto S, Kanno H, Hirose S, Yamamoto T. Reduced PLP1 expression in induced pluripotent stem cells derived from a Pelizaeus-Merzbacher disease patient with a partial PLP1 duplication. J Hum Genet. 2012 Sep;57(9):580-6. doi: 10.1038/jhg.2012.71. Epub 2012 Jun 14. PMID 22695888
- [Background] Stankiewicz P, Beaudet AL. Use of array CGH in the evaluation of dysmorphology, malformations, developmental delay, and idiopathic mental retardation. Curr Opin Genet Dev. 2007 Jun;17(3):182-92. doi: 10.1016/j.gde.2007.04.009. Epub 2007 Apr 30. PMID 17467974
- [Background] Stasia MJ, Mollin M, Martel C, Satre V, Coutton C, Amblard F, Vieville G, van Montfrans JM, Boelens JJ, Veenstra-Knol HE, van Leeuwen K, de Boer M, Brion JP, Roos D. Functional and genetic characterization of two extremely rare cases of Williams-Beuren syndrome associated with chronic granulomatous disease. Eur J Hum Genet. 2013 Oct;21(10):1079-84. doi: 10.1038/ejhg.2012.310. Epub 2013 Jan 23. PMID 23340515
- [Background] Stevenson, R. E., Schwartz, C. E. & Schroer, R. J. X-Linked Mental Retardation. 2000. Oxford Univ. Press
- [Background] Takahashi K, Yamanaka S. Induction of pluripotent stem cells from mouse embryonic and adult fibroblast cultures by defined factors. Cell. 2006 Aug 25;126(4):663-76. doi: 10.1016/j.cell.2006.07.024. Epub 2006 Aug 10. PMID 16904174
- [Background] Thienpont B, de Ravel T, Van Esch H, Van Schoubroeck D, Moerman P, Vermeesch JR, Fryns JP, Froyen G, Lacoste C, Badens C, Devriendt K. Partial duplications of the ATRX gene cause the ATR-X syndrome. Eur J Hum Genet. 2007 Oct;15(10):1094-7. doi: 10.1038/sj.ejhg.5201878. Epub 2007 Jun 20. PMID 17579672
- [Background] Wapinski OL, Vierbuchen T, Qu K, Lee QY, Chanda S, Fuentes DR, Giresi PG, Ng YH, Marro S, Neff NF, Drechsel D, Martynoga B, Castro DS, Webb AE, Sudhof TC, Brunet A, Guillemot F, Chang HY, Wernig M. Hierarchical mechanisms for direct reprogramming of fibroblasts to neurons. Cell. 2013 Oct 24;155(3):621-35. doi: 10.1016/j.cell.2013.09.028. Epub 2013 Oct 24. PMID 24243019
- [Background] Yanaba K, Nakagawa H, Takeda Y, Koyama N, Sugano K. Muir-Torre syndrome caused by partial duplication of MSH2 gene by Alu-mediated nonhomologous recombination. Br J Dermatol. 2008 Jan;158(1):150-6. doi: 10.1111/j.1365-2133.2007.08233.x. Epub 2007 Oct 17. PMID 17941949
- [Background] Yang N, Ng YH, Pang ZP, Sudhof TC, Wernig M. Induced neuronal cells: how to make and define a neuron. Cell Stem Cell. 2011 Dec 2;9(6):517-25. doi: 10.1016/j.stem.2011.11.015. PMID 22136927